CLINICAL TRIAL: NCT03262233
Title: Clinical Relevance of Stress Neuroadaptation in Tobacco Dependence
Brief Title: Stress Neuroadaptation in Tobacco Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017-0433
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Active Deprived (Experimental): 21 mg nicotine patches and 2 mg nicotine lozenges
  + First NPU task takes place 24 hours after start of quit attempt
  Interventions: Combination Product: nicotine
- Active Non-deprived (Experimental): 21 mg nicotine patches and 2 mg nicotine lozenges
  + First NPU task takes place during normal smoking prior to quit attempt
  Interventions: Combination Product: nicotine
- Placebo Deprived (Active Comparator): Placebo patches and placebo lozenges
  + First NPU task takes place 24 hours after start of quit attempt
  Interventions: Other: placebo
- Placebo Non-deprived (Active Comparator): Placebo patches and placebo lozenges
  + First NPU task takes place during normal smoking prior to quit attempt
  Interventions: Other: placebo

INTERVENTIONS:
Combination Product: nicotine
  Arms: Active Deprived; Active Non-deprived
Other: placebo
  Arms: Placebo Deprived; Placebo Non-deprived

SUMMARY:
The objective of the current study is to evaluate the validity of the No Shock, Predictable Shock, Unpredictable Shock (NPU) stressor task for use as a surrogate endpoint to predict short-term clinical outcomes among smokers during a smoking cessation attempt.

DETAILED DESCRIPTION:
Smokers recruited for this study are randomly assigned at a screening session to complete the NPU stressor task pre-quit or post-quit (i.e., nicotine deprived or non-deprived). Participants are also randomized to receive either placebo or active combination nicotine replacement therapy (NRT; patches and lozenges) for a two week smoking cessation period. The NPU stressor task measures stressor reactivity to predictable and unpredictable stressors (i.e., electric shock). Startle potentiation during predictable and unpredictable stressors (relative to no-shock) provides the primary measures of stressor reactivity in this task. Predictable and unpredictable startle potentiation are used to calculate overall stressor reactivity and selective unpredictable stressor reactivity. Further detail on these reactivity measures is provided in the Independent Variables section. Detail on the quantification of startle potentiation is provided at the end of this registration.

Smokers provide three weeks (1 week pre-quit, 2 weeks post-quit) of brief 4x daily, real-time web-survey reports of recent cigarette use, NRT use, and other measures not relevant to this study's purpose on the participants' smartphones. At two weeks post-quit, smokers are scheduled for a laboratory visit where participants provide an additional report via staff interview of any smoking during the two-week smoking cessation period.

The stressor reactivity measures from the NPU task will be tested as predictors of clinical outcome (i.e., continuous abstinence during the two-week cessation period) to evaluate the validity of each as surrogate endpoints for use in research on stress mechanisms in smoking relapse. Deprivation status at the time of the NPU stressor task will be examined as a moderator of the effect of stressor reactivity to determine if the surrogate endpoints predict clinical outcome generally or only as deprivation increases.

ELIGIBILITY:
Inclusion Criteria:

* cigarette use over 10 cigarettes/day for over two years;
* smoking within the first 30 minutes of waking up
* expired air carbon monoxide (CO) level >6 ppm
* self-reported motivation to quit smoking
* and an agreement to respond to ecological momentary assessment prompts (via SMS) throughout the day for three weeks.

Exclusion Criteria:

* Health screening are performed by questionnaire and reviewed by study staff (RA or Research Specialist) to ensure that smokers can safely use the nicotine patch and lozenge. Specifically, smokers will be excluded for FDA contraindications for nicotine replacement therapy (i.e., no uncontrolled hypertension, recent myocardial infarction, diabetes, heart disease, asthma, stomach ulcers).
* All women of child-bearing potential will be required to agree to use an approved method of birth control to prevent pregnancy during the course of the study.
* All participants will report no medical or psychiatric condition that would contraindicate exposure to electric shock.
* Participants with uncorrected auditory or visual problems will be excluded.

Additional Data Exclusions

1. As part of the NPU stressor task, smokers are asked to indicate if the participant "can be shocked in the next 5 seconds" at various points during the task. Responses to these questions are used to verify that the participant understands the cue-shock contingencies. Smokers who answer < 10 out of 14 questions correctly the NPU stressor task during the experimental session will be excluded from all analyses and replaced.
2. Smokers with 20% of cue trials identified as artifact in the NPU task will be excluded from all analyses and replaced.
3. The analysis will NOT exclude smokers who are startle non-responders given that the use of these surrogate endpoints in practice would likely need to include these individuals to avoid unnecessary data loss.
4. Smokers who do not report a complete abstinence between quit date/time and final laboratory visit (which occurs 12-36 hours later) will be considered to not have quit and will be excluded from all analyses and replaced.
5. Smokers for whom the investigators cannot definitively quantify an outcome with respect to continuous abstinence will be excluded from all analyses and replaced. Any report of smoking during the two-week cessation period (reported either during the 4x daily web surveys or the laboratory visit at 2 weeks) is sufficient to code the smoker to have lapsed (i.e., not continuously abstinent), even if the participants do not complete the full two weeks of web surveys and/or the 2-week laboratory visit. However, the status of smokers who report no smoking during the cessation attempt but have both a high level of missing data from the web surveys (> 25% of reports) and no two-week laboratory visit report will be deemed uncertain. These smokers will be excluded and replaced.
6. The investigators will conduct case analyses to identify participants who are model outliers with Bonferroni-corrected studentized residuals p < 0.05. These model outliers will be excluded but NOT replaced (because the participants are not identified until after data collection has been completed).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on the data repository at Open Science Foundation
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be available on submission of first manuscript based on study
Access Criteria: Data are completely open
URL: https://osf.io/dz9yu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Deprived | Active Non-Deprived | Placebo Deprived | Placebo Non-deprived
Started | 53 | 53 | 59 | 61
Completed | 35 | 32 | 34 | 32
Not Completed | 18 | 21 | 25 | 29
Not completed — Withdrawal by Subject | 12 | 8 | 21 | 13
Not completed — Declined due to shock | 1 | 2 | 2 | 3
Not completed — Protocol Violation | 5 | 10 | 2 | 13
Not completed — data collection artifact | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Deprived | Active Non-Deprived | Placebo Deprived | Placebo Non-Deprived | Total
Number analyzed (Participants) | 35 | 32 | 34 | 32 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (10.7) | 39.7 (12.4) | 40.6 (12.3) | 42 (11.3) | 40 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 12 | 11 | 50
  Male | 21 | 19 | 22 | 21 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 34 | 32 | 33 | 32 | 131
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 1 | 3
  Asian | 0 | 01 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 7 | 11 | 9 | 36
  White | 26 | 21 | 21 | 21 | 89
  More than one race | 0 | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 32 | 34 | 32 | 133

OUTCOME MEASURES:

1. Primary Outcome: Overall Stressor Reactivity
Description: The average of unpredictable startle potentiation and predictable startle potentiation during the first administration of the NPU stressor task.
Time Frame: up to 24 hours after start of cessation attempt (deprived groups); during normal smoking prior to quit attempt, ie. Baseline (non-deprived groups)
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Active Deprived | Active Non-deprived | Placebo Deprived | Placebo Non-deprived
Number analyzed (Participants) | 35 | 32 | 34 | 32
microvolts | 25.1 (23.0) | 22.5 (24.4) | 32.3 (29.6) | 16.9 (17.7)

2. Primary Outcome: Relative Unpredictable Stressor Reactivity
Description: Unpredictable startle potentiation minus predictable startle potentiation during the first administration of the NPU stressor task
Time Frame: up to 24 hours post cessation attempt (deprived groups); during normal smoking prior to quit attempt, ie. Baseline (non-deprived groups)
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Active Deprived | Active Non-Deprived | Placebo Deprived | Placebo Non-deprived
Number analyzed (Participants) | 35 | 32 | 34 | 32
microvolts | -6.77 (14.0) | -7.91 (14.4) | -6.06 (12.3) | -4.99 (14.0)

3. Primary Outcome: Change in Overall Stressor Reactivity
Description: A difference score of overall stressor reactivity during the second administration of the NPU stressor task relative to the first NPU stressor task
Time Frame: baseline and up to 14 days post cessation attempt (non-deprived groups); baseline and up to 24 hours post quit attempt (deprived groups)
Measure: Mean (Standard Deviation); unit: change in microvolts
Arm/Group | Active Deprived | Active Non-Deprived | Placebo Deprived | Placebo Non-deprived
Number analyzed (Participants) | 35 | 32 | 34 | 32
change in microvolts | -2.94 (16.3) | 0.929 (13.0) | -10.3 (24.0) | 4.78 (13.6)

4. Primary Outcome: Change in Relative Unpredictable Stressor Reactivity
Description: A difference score of relative unpredictable stressor reactivity during the second administration of the NPU stressor task relative to the first NPU stressor task
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: change in microvolts
Arm/Group | Active Deprived | Active Non-Deprived | Placebo Deprived | Placebo Non-deprived
Number analyzed (Participants) | 35 | 32 | 34 | 32
change in microvolts | 1.95 (15.5) | 3.99 (14.8) | 0.889 (16.0) | -1.35 (11.3)

ADVERSE EVENTS:
Time Frame: through 14 days post quit
Arm/Group | Active Deprived | Active Non-deprived | Placebo Deprived | Placebo Non-deprived
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/32 | 0/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/32 | 0/34 | 0/32
Other Adverse Events (participants affected / at risk) | 0/35 | 0/32 | 0/34 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT03262233/Prot_SAP_000.pdf